CLINICAL TRIAL: NCT04620967
Title: Fast-Acting Insulin Aspart and Insulin Pump Settings: THE FAST PUMP SETTING STUDY
Brief Title: Fast-Acting Insulin Aspart and Insulin Pump Settings
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kirsten Nørgaard (Other)
Responsible Party: Sponsor-Investigator, Kirsten Nørgaard, Senior Consultant, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-001158-23; H-20022359 (Other: Scientific Ethical Committee of the Capital Region of Denmark)
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Type 1 Diabetes
Keywords: Insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, cross-over study with two 16-week intervention periods separated by a 3-week washout period comparing Fiasp with Iasp in adults with type 1 diabetes treated with insulin pump and CGM.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Group allocation is concealed to participants as well as investigators until all participants have completed the study. The allocation for a participant may be revealed in a medical emergency if knowledge about the treatment allocation would influence the treatment of the person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iasp-Fiasp (Experimental): First period: Insulin pump with Iasp Second period: Insulin pump with Fiasp
  Interventions: Drug: Insulin aspart; Drug: Fast-acting insulin aspart
- Fiasp-Iasp (Experimental): First period: Insulin pump with Fiasp Second period: Insulin pump with Iasp
  Interventions: Drug: Insulin aspart; Drug: Fast-acting insulin aspart

INTERVENTIONS:
Drug: Insulin aspart — Insulin aspart (Iasp) in insulin pump
Drug: Fast-acting insulin aspart — Fast-acting insulin aspart (Fiasp) in insulin pump

SUMMARY:
To clarify the role of fast-acting insulin aspart (Fiasp) in insulin pump-treated type 1 diabetes more research is needed.

The aim of this study is twofold:

1. to compare the effects of Fiasp and Iasp in adults with type 1 diabetes who are using insulin pump and CGM and who are attending a diabetes out-patient clinic with extensive expertise in insulin pump and CGM therapy.
2. to determine differences in insulin pump settings when insulin pumps are optimally adjusted to each of the two insulin types.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for ≥ 5 years
* HbA1c 53-75 mmol/mol (7.0-9.0%)
* Insulin pump treatment for ≥ 6 months (all insulin pump makes except hybrid closed-loop systems are eligible for inclusion)
* CGM use for ≥ 6 months (all CGM makes are eligible for inclusion)
* Carbohydrate counting for all snacks and meals
* Use of the insulin pump bolus calculator for all meals and snacks

Exclusion Criteria:

* Breast-feeding, pregnant, planning to become pregnant or of child-bearing potential and not using adequate contraceptive methods
* Gastroparesis (clinical assessment)
* Shift work
* Changing insulin needs throughout the menstrual cycle that requires different basal rate patterns
* Use of a hybrid closed-loop system
* Use of flash glucose monitoring
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Chronic paracetamol use
* Alcohol or drug abuse
* Severe cardiac disease or retinopathy contraindicating HbA1c below 53 mmol/mol
* Impaired renal function (eGFR< 60 ml/min/1.73 m2)
* History of local skin reactions to Fiasp and/or Iasp
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation
* Lack of compliance with key study procedures at the discretion of the investigator
* Unacceptable adverse events at the discretion of the investigator
* Less than 40 weeks guarantee remaining on insulin pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Time in range | Last two weeks of the 16-week interventions
  Difference in time spent with glucose values in the range 3.9-10.0 mmol/l between Fiasp and Iasp treatment assessed by continuous glucose monitoring

SECONDARY OUTCOMES:
Mean glucose | Last two weeks of the 16-week interventions
  Difference in mean glucose between Fiasp and Iasp treatment assessed by continuous glucose monitoring
Coefficient of variation | Last two weeks of the 16-week interventions
  Difference in coefficient of variation between Fiasp and Iasp treatment assessed by continuous glucose monitoring
Time below range level 1 | Last two weeks of the 16-week interventions
  Difference in time spent with glucose values below 3.9 mmol/l between Fiasp and Iasp treatment assessed by continuous glucose monitoring
Time below range level 2 | Last two weeks of the 16-week interventions
  Difference in time spent with glucose values below 3.0 mmol/l between Fiasp and Iasp treatment assessed by continuous glucose monitoring
Time above range level 1 | Last two weeks of the 16-week interventions
  Difference in time spent with glucose values above 10.0 mmol/l between Fiasp and Iasp treatment assessed by continuous glucose monitoring
Time above range level 2 | Last two weeks of the 16-week interventions
  Difference in time spent with glucose values above 13.9 mmol/l between Fiasp and Iasp treatment assessed by continuous glucose monitoring
Fructosamine | 16 weeks
  Difference in change in fructosamine between Fiasp and Iasp treatment
Total daily insulin dose | Last two weeks of the 16-week interventions
  Difference between Fiasp and Iasp treatment in total daily insulin dose
Total daily basal insulin dose | Last two weeks of the 16-week interventions
  Difference between Fiasp and Iasp treatment in total daily basal insulin dose
Total daily bolus insulin dose | Last two weeks of the 16-week interventions
  Difference between Fiasp and Iasp treatment in total daily bolus insulin dose
Severe hypoglycemia | 16 weeks
  Difference between Fiasp and Iasp treatment in number of severe hypoglycemia events
Ketoacidosis | 16 weeks
  Difference between Fiasp and Iasp treatment in number of ketoacidosis events

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nørgaard, MD DMSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark